CLINICAL TRIAL: NCT03925779
Title: Dexmedetomidine Versus Propofol-Remifentanil Conscious Sedation for Outpatient Colonoscopy: A Prospective Randomized Double-blind Trial.
Brief Title: Conscious Sedation for Outpatient Colonoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Abd-Elazeem Abd-Elhameed Elbakry, Associate professor of anaesthesia, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2019/3/15/9
Record Dates: First submitted 2019-04-21; First posted 2019-04-24 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Conscious Sedation
MeSH Terms: interventions — Dexmedetomidine; Propofol; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: A blinded investigator that was not involved in the anaesthetic management of the patients, collected the intra-operative and postoperative data. The patients and colonoscopist were blinded to group allocation. For blinding purposes, two drug infusion pumps were used in every patient where the infusion pumps and i.v. connection lines were concealed to avoid identification.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Dexmedetomidine)Dex group (Active Comparator): The patients will be administered a loading dose of i.v. dexmedetomidine 1 μg/kg over 10 min, followed by a continuous infusion of 0.2-1 μg/kg/h, titrated according to the sedation score, till the end of the procedure
  Interventions: Drug: Dexmedetomidine
- Propofol-Remifentanil (P-R) group (Active Comparator): Propofol will be started by a loading dose of 0.5 mg/kg over 3-5 minutes then a maintenance infusion of 25-75 μg kg/min. Remifentanil infusion will be started at 1 μg kg over one minute then and 0.01-0.1 μg kg/min.
  Interventions: Drug: Propofol; Drug: Remifentanil

INTERVENTIONS:
Drug: Dexmedetomidine — dexmedetomidine sedation
  Other Names: dexmedetomidine infusion
  Arms: (Dexmedetomidine)Dex group
Drug: Propofol — propofol sedation
  Other Names: propofol infusion
  Arms: Propofol-Remifentanil (P-R) group
Drug: Remifentanil — Remifentanil sedation
  Other Names: Remifentanil infusion
  Arms: Propofol-Remifentanil (P-R) group

SUMMARY:
Although colonoscopy is a mildly painful procedure, the pain and the procedure itself are distressful for most patients. This raises the attention for using different sedation regimens aiming at maintaining optimal sedation level with maintained airway and stable haemodynamics all through the procedure. The present study was scheduled to investigate the sedative efficacy of dexmedetomedine versus propofol-remifentanil for outpatient colonoscopy.

DETAILED DESCRIPTION:
Eighty patients undergoing outpatient colonoscopy will be randomized into two equal groups. In Dexmedetomidine (DEX) group the patients will be administered a loading dose of i.v. dexmedetomidine 1 μg/kg over 10 min, followed by a continuous infusion of 0.2-1 μg/kg/h, titrated according to the sedation score, till the end of the procedure. In the PR group, propofol will be started by a loading dose of 0.5 mg/kg over 3-5 minutes then a maintenance infusion of 25-75 μg kg/min. Remifentanil infusion will be started at 1 μg kg over one minute then and 0.01-0.1 μg kg/min. If the patient complained of pain or discomfort, the infusion rates of dexmedetomidine (DEX group) or propofol-remifentanil (P-R group) will be increased. If the higher limit of the dose range of the study drugs reached, additional fentanyl 0.5 μg/kg i.v. boluses will be administered. Rescue medication consisting of propofol boluses of 0.5 mg/kg i.v. will be given if the previous protocol failed. Sedation score,haemodynamics, end-tidal carbon dioxide, oxygen saturation, total fentanyl, propofol bolus doses, patient and colonoscopist satisfaction and side effects will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II physical status
* 18-65 years
* Scheduled for elective colonoscopy

Exclusion Criteria:

* History of allergy to any of the study drugs
* Alcohol or drug abuse.
* Second and third-degree heart block.
* Morbid obesity.
* Pregnant and lactating women.
* Psychiatric disorders.
* Severe cardiac, respiratory, renal, and liver diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
Sedation | Perioperative
  Degree of sedation by Ramsay sedation score from 1 inadequate sedation to 6 excessive sedation.

SECONDARY OUTCOMES:
Mean arterial blood pressure | Perioperative
  Mean arterial blood pressure in mmHg
Heart rate | Perioperative
  Heart rate in beats/minutes
Oxygen saturation | Perioperative
  Arterial oxygen saturation as a percentage of the total haemoglobin.
Hypotension | Perioperative
  Number of patients with hypotension
Bradycardia | Perioperative
  Number of patients with bradycardia
Analgesia | Perioperative
  Measured by visual analogue scale [from 0 "no pain" to 10 "worst imaginable pain"]

CONTACTS AND LOCATIONS:
Overall Officials: Abd-Elazeem A Elbakry, MD, Principal Investigator — Associate professor
Locations (1):
- Faculty of Medicine, Cairo, Shebin El-kom, Egypt